CLINICAL TRIAL: NCT04526444
Title: E-health Interventions to Promote Physical Activity Among Inactive Adults: a Hybrid Type I Effectiveness-implementation Randomized Controlled Trial
Brief Title: E-health Interventions to Promote Physical Activity Among Inactive Adults
Acronym: ONWARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: UiT The Arctic University of Norway (Other); SINTEF Health Research (Other); PAI Health Norway AS (Unknown); St. Olavs Hospital (Other); Norwegian University of Science and Technology (Other); Frisklivssentralen (Unknown); Laval University (Other); Les Mills International (Unknown)
Responsible Party: Principal Investigator, Paolo Zanaboni, Senior researcher, University Hospital of North Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 66573
Record Dates: First submitted 2020-08-07; First posted 2020-08-25 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Physical Activity Promotion Among Inactive Adults
MeSH Terms: interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ftiness tracker (Experimental): Participants in the group A will be provided the fitness tracker Mi Smart Band 5 with the computational algorithm PAI.
  Interventions: Device: Fitness tracker
- Home training platform and fitness tracker (Experimental): Participants in group B will be provided with both the fitness tracker Mi Smart Band 5 with the computational algorithm PAI and access to Les Mills On Demand to perform training classes from home.
  Interventions: Device: Fitness tracker; Other: Online training
- Peer support, home training platform and fitness tracker and (Experimental): Participants in group C will be offered the fitness tracker Mi Smart Band 5 with the computational algorithm PAI, Les Mills On Demand and additional peer support via social media.
  Interventions: Device: Fitness tracker; Other: Online training; Other: Peer support via social media

INTERVENTIONS:
Device: Fitness tracker — Fitness tracker Mi Smart Band 5 with the computational algorithm PAI
Other: Online training — Les Mills On Demand
  Arms: Home training platform and fitness tracker; Peer support, home training platform and fitness tracker and
Other: Peer support via social media — Facebook group
  Arms: Peer support, home training platform and fitness tracker and

SUMMARY:
The project addresses physical inactivity as a global health issue. Physical inactivity is the fourth leading risk factor for global mortality. Moreover, inactive adults have a higher risk to develop lifestyle diseases. To date, there is preliminary evidence of the efficacy in the use of certain strategies including fitness technologies and digital interventions for physical activity (PA) promotion. Intervention studies are needed to test the effectiveness of PA promotion strategies.

A Hybrid Type I effectiveness-implementation randomised controlled trial (RCT) will investigate the effects of 1) fitness trackers, 2) home-based online training, and 3) peer support via social media among inactive adults. The design will allow testing the study outcomes while gathering information on implementation in a real-world situation. The study will produce evidence on whether these interventions increase the levels of PA among inactive adults and improve health outcomes. Increased PA will also result in better primary prevention of lifestyle diseases.

ELIGIBILITY:
Inclusion Criteria:

* young (18-40 years) or middle aged (40-55 years) healthy adults, both men and women;
* inactive (undertaking less than 150 min of moderate-intensity PA per week) in the last 3 months;
* living in the Troms and Finnmark county;
* current owner of a smartphone;
* able to understand training instructions in English language.

Exclusion Criteria:

* presence of disabilities which might reduce the ability to perform exercise;
* presence of conditions which might prevent from safely exercise;
* lack of Internet connection at home;
* lack of space to exercise safely at home (recommended 4 sqm).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Level of physical activity short-term | 6 months
  Time spent in moderate to vigorous physical activity
Level of physical activity medium-term | 12 months
  Time spent in moderate to vigorous physical activity
Level of physical activity long-term | 18 months
  Time spent in moderate to vigorous physical activity

SECONDARY OUTCOMES:
Adherence to recommendation short-term | 6 months
  Proportion of participants reaching the recommendation for physical activity
Adherence to recommendation medium-term | 12 months
  Proportion of participants reaching the recommendation for physical activity
Adherence to recommendation long-term | 18 months
  Proportion of participants reaching the recommendation for physical activity
Physical fitness short-term | 6 months
  VO2 max (estimated)
Physical fitness medium-term | 12 months
  VO2 max (estimated)
Physical fitness long-term | 18 months
  VO2 max (estimated)
Body Mass Index (BMI) short-term | 6 months
Body Mass Index (BMI) medium-term | 12 months
Body Mass Index (BMI) long-term | 18 months
Waist circumference short-term | 6 months
Waist circumference medium-term | 12 months
Waist circumference long-term | 18 months
EQ-5D-5L (EuroQol 5 Dimension 5 Level) Quality of life short-term | 6 months
  EQ-5D-5L has 5 dimensions and 5 levels from 1 to 5 in each dimension (1 is no problems). It also includes a Visual Analogue scale from 0 to 100 (100 is best possible health). Rating can be transformed to a score with min -0.654 and max (1 is no problems in all dimensions).
EQ-5D-5L (EuroQol 5 Dimension 5 Level) Quality of life medium-term | 12 months
  EQ-5D-5L has 5 dimensions and 5 levels from 1 to 5 in each dimension (1 is no problems). It also includes a Visual Analogue scale from 0 to 100 (100 is best possible health). Rating can be transformed to a score with min -0.654 and max (1 is no problems in all dimensions).
EQ-5D-5L (EuroQol 5 Dimension 5 Level) Quality of life long-term | 18 months
  EQ-5D-5L has 5 dimensions and 5 levels from 1 to 5 in each dimension (1 is no problems). It also includes a Visual Analogue scale from 0 to 100 (100 is best possible health). Rating can be transformed to a score with min -0.654 and max (1 is no problems in all dimensions).
Perceived competence for exercise (PCS-EX) short-term | 6 months
  4 items. Min 4, max 28 (28 high competence)
Perceived competence for exercise (PCS-EX) medium-term | 12 months
  4 items. Min 4, max 28 (28 high competence)
Perceived competence for exercise (PCS-EX) long-term | 18 months
  4 items. Min 4, max 28 (28 high competence)
Self-efficacy for exercise (SEE) Scale short-term | 6 months
  Scale with 9 items, min 0 and max 90. Higher score indicates higher self-efficacy for exercise.
Self-efficacy for exercise (SEE) Scale medium-term | 12 months
  Scale with 9 items, min 0 and max 90. Higher score indicates higher self-efficacy for exercise.
Self-efficacy for exercise (SEE) Scale long-term | 18 months
  Scale with 9 items, min 0 and max 90. Higher score indicates higher self-efficacy for exercise.
Social Support (SSES) short-term | 6 months
  13 items answered two times, one for family and one for friends. Min 13, max 65 (65 highest level of social support)
Social Support (SSES) medium-term | 12 months
  13 items answered two times, one for family and one for friends. Min 13, max 65 (65 highest level of social support)
Social Support and Exercise scale (SSES) long-term | 18 months
  13 items answered two times, one for family and one for friends. Min 13, max 65 (65 highest level of social support)
Reasons for performing physical activity short-term | 6 months
  Behavioural Regulation Exercise Questionnaire (BREQ-2).
Reasons for performing physical activity medium-term | 12 months
  Behavioural Regulation Exercise Questionnaire (BREQ-2).
Reasons for performing physical activity long-term | 18 months
  Behavioural Regulation Exercise Questionnaire (BREQ-2).
System Usability Scale (SUS) | 6 months
  10 items, min 0 max 100 (above 68 is above the average).
Users' perspectives on intervention through interviews short-term | 6 months
  Qualitative data derived from semi-structured interviews with participants.
Users' perspectives on intervention through interviews long-term | 18 months
  Qualitative data derived from semi-structured interviews with participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian Centre for E-health Research, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sagelv EH, Manskow US, Antypas K, Morseth B, Aamot Aksetoy IL, Nes BM, Gagnon MP, Zanaboni P. Online interventions to increase physical activity levels in self-reported inactive adults: the ONWARDS randomised controlled trial. BMJ Open Sport Exerc Med. 2025 Jun 16;11(2):e001816. doi: 10.1136/bmjsem-2023-001816. eCollection 2025. PMID 40546750
- [Derived] Manskow US, Sagelv EH, Antypas K, Zanaboni P. Adoption, acceptability and sustained use of digital interventions to promote physical activity among inactive adults: a mixed-method study. Front Public Health. 2024 Jan 4;11:1297844. doi: 10.3389/fpubh.2023.1297844. eCollection 2023. PMID 38239801
- [Derived] Zanaboni P, Manskow US, Sagelv EH, Morseth B, Edvardsen AE, Aamot IL, Nes BM, Hastings B, Gagnon MP, Antypas K. Digital interventions to promote physical activity among inactive adults: A study protocol for a hybrid type I effectiveness-implementation randomized controlled trial. Front Public Health. 2022 Oct 21;10:925484. doi: 10.3389/fpubh.2022.925484. eCollection 2022. PMID 36339169